CLINICAL TRIAL: NCT06483139
Title: The Effect of Novel Treatments in Improving Renal Outcomes Among Patients With Light Chain Cast Nephropathy
Brief Title: Novel Treatments in Improving Renal Outcomes in Light Chain Cast Nephropathy
Status: Recruiting | Type: Observational
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Janssen, LP (Industry); Baystate Health (Other); Boston Medical Center (Other); Dana-Farber Cancer Institute (Other); Massachusetts General Hospital (Other); Mayo Clinic (Other); M.D. Anderson Cancer Center (Other); Medical University of South Carolina (Other); H. Lee Moffitt Cancer Center and Research Institute (Other); Icahn School of Medicine at Mount Sinai (Other); Northwell Health (Other); Ochsner Health System (Other); Ohio State University (Other); Stanford University (Other); Texas Medical Center (Unknown); Thomas Jefferson University (Other); University of Alabama at Birmingham (Other); University of California, Los Angeles (Other); University of Chicago (Other); University of Colorado Health (Other); University of Minnesota (Other); University of New Mexico (Other); University of Pennsylvania (Other); University of Pittsburgh (Other); University of Virginia (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Shruti Gupta, Associate Physician, Director of Onconephrology, Brigham and Women's Hospital
Other Study IDs: 2021P002205
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Multiple Myeloma; Light Chain Nephropathy; Acute Kidney Injury
MeSH Terms: conditions — Multiple Myeloma; Acute Kidney Injury | interventions — Plasma Exchange; daratumumab

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (4):
- Patients treated with plasma exchange: Treated with plasma exchange ithin 30 days of diagnosis of light chain cast nephropathy
  Interventions: Procedure: Plasma exchange
- Patients not treated with plasma exchange: Patients not treated with plasma exchange within 30 days of diagnosis of light chain cast nephropathy
- Patients treated with daratumumab: Patients treated with daratumumab within 30 days of diagnosis of light chain cast nephropathy
  Interventions: Drug: Daratumumab
- Patients not treated with daratumumab: Patients treated with daratumumab within 30 days of diagnosis of light chain cast nephropathy

INTERVENTIONS:
Procedure: Plasma exchange — Patients treated with plasma exchange within 30 days of diagnosis of light chain cast nephropathy Patients not treated with daratumumab within 30 days of diagnosis of light chain cast nephropathy
  Groups: Patients treated with plasma exchange
Drug: Daratumumab — Patients treated with daratumumab within 30 days of diagnosis of light chain cast nephropathy
  Groups: Patients treated with daratumumab

SUMMARY:
Objective 1: To test whether treatment with plasma exchange improves renal recovery in patients with light chain cast nephropathy Objective 2: To compare renal outcomes among patients treated with plasma exchange versus daratumumab-based regimens versus non-daratumumab based-regimens.

DETAILED DESCRIPTION:
Objective 1:

We will collect data from patients treated with plasma exchange from major centers across the United States to investigate whether plasma exchange improves renal outcomes.

Specifically, we will collect data on at least 150 patients treated with plasma exchange along with 300 control patients not treated with plasma exchange.

Objective 2:

We will compare renal outcomes among patients with light chain cast nephropathy and AKI treated with plasma exchange (n=150) versus daratumumab based regimen (eg Dara-CyborD) (n=150) versus other novel regimens (e.g., CyborD or another non-daratumumab-based regimen) (n=150). We will examine whether patients who receive dara-based regimens are more likely to have renal recovery compared to patients who do not receive dara-based regimens and to patients who receive plasma exchange. Given the infrequency with which plasma exchange is performed on a single-center level, we will compare outcomes among patients treated with plasma exchange, utilizing data from the multicenter study to those patients who were treated with daratumumab-based regimens without plasma exchange versus non- daratumumab-based regimen.

ELIGIBILITY:
Inclusion Criteria for Plasma Exchange-Treated Patients:

1. Adult (≥18 years old)
2. Either a new diagnosis of multiple myeloma confirmed by bone marrow plasmayctosis >10% or acute relapse of multiple myeloma
3. Light chain cast nephropathy, with involved light chain >500 mg/L
4. Acute kidney injury, defined as ≥1.5-fold rise in SCr from baseline (as defined in study outcomes) or the need for renal replacement therapy (RRT).
5. Treated with at least 1 round of plasma exchange within 30 days of diagnosis of cast nephropathy
6. Treated with plasma exchange in 2010 or later

Inclusion Criteria for Control Patients:

1. Adult (≥18 years old)
2. Either a new diagnosis of multiple myeloma confirmed by bone marrow plasmayctosis >10% or acute relapse of multiple myeloma
3. Light chain cast nephropathy, with involved light chain >500 mg/L
4. Acute kidney injury, defined as ≥1.5-fold rise in SCr from baseline or the need for renal replacement therapy (RRT)

Exclusion Criteria for Both Plasma Exchange-Treated Patients and Control Patients:

1. Patients with end stage kidney disease
2. Patients with amyloidosis or monoclonal immunoglobulin deposition disease
3. Patients with chronic lymphocytic leukemia, plasma cell leukemia, or Waldenstrom's
4. Moribund condition (e.g., patients who died within 48 hours of initiation of plasma exchange)
5. Active urinary tract obstruction on renal imaging
6. Patients with significant albuminuria (≥2+ on urinary dipstick or >10% fraction on UPEP)
7. Patients with other biopsy-proven causes of AKI (non-cast nephropathy lesions)
8. Patients who did not receive clone-directed therapy for myeloma
9. Patients who received plasma exchange >30 days from the time of diagnosis of cast nephropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with multiple myeloma and clinically-suspected or biopsy-proven light chain cast nephropathy
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
The primary composite outcome is the rate of survival with renal recovery within 90 days from the diagnosis of light chain cast nephropathy. | 90 days
  To meet the primary outcome, patients must be alive, not RRT-dependent (e.g., were never on dialysis/no longer on dialysis), and have a decline of at least one stage of AKI severity compared to their highest AKI stage achieved at the time of light chain cast nephropathy-associated AKI. AKI staging will be based on the Kidney Disease Improving Global Outcomes (KDIGO) criteria, where stage 1 is a 1.5-1.9-fold rise in SCr from baseline; stage 2 is a 2-2.9-fold rise from baseline; and stage 3 is a 3-fold rise in SCr from baseline or initiation of RRT. Baseline SCr is defined as the lowest SCr in the 365 days preceding the diagnosis of light chain cast nephropathy.

SECONDARY OUTCOMES:
The proportion of patients with Receipt of RRT within 30 days, 60 days, and 90 days following diagnosis of light chain cast nephropathy | 30, 60, 90 days
  The proportion of patients with Receipt of RRT within 30 days, 60 days, and 90 days following diagnsosis of LCCN
The proportion of patients with Progressive AKI | 30, 60, 90 days
  Defined as progression from existing AKI (stage 2) to a higher stage (stage 3 or receipt of RRT) within 30, 60, and 90 days following diagnosis of light chain cast nephropathy. AKI staging at each of these time points will be defined based on KDIGO criteria outlined above.
Survival to hospital discharge | 30 days
  Survival to hospital discharge and KRT-independent among patients admitted within 30 days of the diagnosis of light chain cast nephropathy.
Renal function (SCr) at hospital discharge | 30 days
  Renal function (SCr) at hospital discharge (% increase compared to baseline) among patients who are admitted within 30 days of their diagnosis of light chain cast nephropathy
Time to first renal recovery | 180 days
  Renal recovery will be defined as not RRT-dependent, and with nadir SCr returning to <50% of baseline. This will be assessed within 180 days following the diagnosis of light chain cast nephropathy
Kidney recovery | 30 (+/-15), 60 (+/-15), 90 (+/-30) days, and 180 days (+/-60 days)
  at 30 (+/-15), 60 (+/-15), 90 (+/-30) days, and 180 days (+/-60 days) following the diagnosis of light chain cast nephropathy, , defined as survival, KRT-independent, and with SCr <1.5-fold baseline at each of the above time points.
Overall survival at day 90, 180, 360, with day 0 defined as date of LCCN diagnosis. Patients who die within 48 hours of the diagnosis will be excluded. | 90, 180, 360 days
  At day 90, 180, 360, with day 0 defined as date of LCCN diagnosis
Adverse events | 60 days
  Infection, re-hospitalization, transfusion reactions, bleeding diatheses.

CONTACTS AND LOCATIONS:
Overall Officials: Shruti Gupta, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No